CLINICAL TRIAL: NCT07103096
Title: Infiltration in Rheumatology With 3D Virtual Reality Headset Pilot Study for the Evaluation of Satisfaction and Feasibility According to Location (Icare)
Brief Title: Infiltration in Rheumatology With 3D Virtual Reality Headset Pilot Study for the Evaluation of Satisfaction (ICARE)
Acronym: Icare
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250404; IDRCB 2025-A00458-41 (Other: ANSM)
Record Dates: First submitted 2025-05-14; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Infiltration
Keywords: infiltration; 3D virtual reality headset

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infiltration: Patient requiring infiltration of the spine (high epidural or sacrococcygeal hiatus) of the subacromial-deltoid bursa or the knee

SUMMARY:
This study is to evaluate the satisfaction and feasibility according to the location of the use of a 3D virtual reality headset during an infiltration in rheumatology.

DETAILED DESCRIPTION:
The performance of infiltrative procedures in rheumatology is common, even daily, practice. It may be associated with anticipatory anxiety and pain (for example, during a shoulder infiltration, there is a significant difference between anticipated pain and pain felt with a visual analogue scale of 6.03 versus 3.17, P < 0.001) as well as pain and anxiety during the procedure. Certain techniques are used to limit this anxiety and pain in common practice such as explaining the procedure before and during its performance, the atmosphere (particularly musical atmosphere) and decoration of the room where the procedure takes place (relaxing images visible to the patient, brightness, people present) and the attitude of the practitioner. More recently, hypnosis and/or 3D virtual reality techniques using a virtual reality headset have been implemented in medicine and particularly in rheumatology to help manage chronic or acute pain. Thus, we currently use a virtual reality headset associated with hypnotic induction (using an audio headset) for the performance of many infiltrative procedures. However, there is no data concerning the acceptability and satisfaction of the patient and the physician of the addition of this technique (VR headset with hypnotic induction) nor its feasibility in current practice (extension of the procedure time for example), during an infiltration nor to know if these data can vary according to the infiltrated location.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patient requiring infiltration of the spine (high epidural or sacrococcygeal hiatus) of the subacromial-deltoid bursa or the knee, regardless of the product infiltrated
* Within the Rheumatology department of Saint-Antoine hospital (consultation or hospitalized)

Exclusion Criteria:

* History of severe psychiatric disorders - History of epilepsy
* Cognitive disorders
* Language barrier - Hearing aid-assisted deafness and/or ophthalmological problems leading to a major loss of vision (advanced cataract, visual impairment)
* Infiltration of the spine (high epidural or sacrococcygeal hiatus), subacromial-deltoid bursa or knee < 6 months
* Characterized depressive disorder diagnosed recently (for less than 6 months) or not stabilized
* Previous use of a virtual reality headset during treatment
* Being under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient requiring infiltration of the spine (high epidural or sacrococcygeal hiatus) of the subacromial-deltoid bursa or the knee
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To assess patient satisfaction with the use of 3D virtual reality with hypnotic induction during infiltration using Modified Client satisfaction score (CSQ-8) | day one
  Modified Client satisfaction score (CSQ-8) Minimum value: 0= not satisfied. Maximum value= 4 totally satisfied. Higher score mean better outcome.

SECONDARY OUTCOMES:
To assess investigator satisfaction | Day one
  Number of times the doctor is satisfied according to the 5-point Likert scale of satisfaction. Minimum value: 0= not satisfied. Maximum value= 5 totally satisfied. Higher score mean better outcome.
To Modified Client satisfaction score (CSQ-8) score according to the location of the infiltration | Day one
  Modified Client satisfaction score (CSQ-8) according to the location of the infiltration. Minimum value: 0= not satisfied. Maximum value= 4 totally satisfied. Higher score mean better outcome.
Assess the patient's anxiety during infiltration using a numerical scale | day one
  Numerical scale patient anxiety during infiltration: mean (standard deviation). Minimum value: 0= Not at all anxious. Maximum value= 10 very anxious. Higher score mean worse outcome.
To Assess the patient's pain during the infiltration using a numerical scale. | day one
  Patient pain numerical scale during infiltration: mean (standard deviation) Minimum value: 0= no pain. Maximum value= 10 the worst pain imaginable. Higher score mean worse outcome.
To Compare pain during infiltration to anticipated pain from infiltration using a numerical scale | day one
  * Numerical scale of pain during infiltration Minimum value: 0= no pain. Maximum value= 10 the worst pain imaginable. Higher score mean worse outcome.
  * Numerical scale of anticipated pain of infiltration. Minimum value: 0= no anticipated pain. Maximum value= 10 the worst anticipated pain imaginable. Higher score mean worse outcome.
Evaluate the added duration of the gesture by using the virtual reality headset | day one
  Duration of the gesture in minutes
Compare the duration of the gesture with hypnotic 3D virtual reality versus the assumed duration without the use of the headset | day one
  Average added time by the Virtual Reality headset according to the doctor
Describe the tolerance of the Virtual Reality headset | day one
  Proportion of immediate side effects to the virtual reality headset

CONTACTS AND LOCATIONS:
Overall Officials: Alice COURTIES, Medical doctor, Principal Investigator — APHP
Locations (1):
- Rheumatology department Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No